CLINICAL TRIAL: NCT01412320
Title: The Impact of Dietary Flavanols on Cardiovascular Dysfunction in End-stage Renal Disease
Brief Title: Cocoa Flavanols in Renal Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Klinik für Kardiologie, Pneumologie und Angiologie (Other)
Responsible Party: Sponsor-Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Christos Rammos, MD Clinic for Cardiology, Pneumology and Angiology, Heinrich-Heine University, Duesseldorf
Organization: Heinrich-Heine University, Duesseldorf (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ESRD_2010
Record Dates: First submitted 2011-08-05; First posted 2011-08-09 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: End Stage Renal Disease; Endothelial Dysfunction
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Chocolate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Flavanol rich cocoa (Experimental)
  Interventions: Other: Cocoa
- Flavanol poor (Experimental)
  Interventions: Other: Cocoa

INTERVENTIONS:
Other: Cocoa — dissolved in water twice daily
  Arms: Flavanol rich cocoa
Other: Cocoa — dissolved in water twice daily
  Arms: Flavanol poor

SUMMARY:
Purpose of the study is to characterize the potential acute and long-term improvement of dietary flavanols on vascular function in patients with end-stage renal disease (ESRD).

Patients will twice daily receive either a flavanol-poor or a flavanol-rich drink. In a double blind, placebo-controlled crossover study the safety, efficacy and acute beneficial effects of flavanol ingestion will be assessed in 10 patients with ESRD. In a 30 day long-term, double blind, placebo-controlled parallel study the chronic effects of dietary flavanols on vascular function in 52 patients with ESRD will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* end stage renal disease
* >18 years
* chronic intermittent hemodialysis

Exclusion Criteria:

* acute Infection
* acute renal failure
* heart failure (NYHA IV)
* pregnancy
* anuria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The effect of flavanols on endothelial function as measured by flow-mediated dilation (FMD) after forearm ischemia and reperfusion. | 30 days
  To study the effect of flavanols on flow mediated dilation of the brachial artery after 5 minutes of forearm ischemia and reperfusion in patients with ESRD

CONTACTS AND LOCATIONS:
Locations (1):
- Heinrich-Heine-University, Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Balzer J, Rassaf T, Heiss C, Kleinbongard P, Lauer T, Merx M, Heussen N, Gross HB, Keen CL, Schroeter H, Kelm M. Sustained benefits in vascular function through flavanol-containing cocoa in medicated diabetic patients a double-masked, randomized, controlled trial. J Am Coll Cardiol. 2008 Jun 3;51(22):2141-9. doi: 10.1016/j.jacc.2008.01.059. PMID 18510961
- [Derived] Colombijn JM, Hooft L, Jun M, Webster AC, Bots ML, Verhaar MC, Vernooij RW. Antioxidants for adults with chronic kidney disease. Cochrane Database Syst Rev. 2023 Nov 2;11(11):CD008176. doi: 10.1002/14651858.CD008176.pub3. PMID 37916745
- [Derived] Luedike P, Rammos C, Pohl J, Heisler M, Totzeck M, Kleophas W, Hetzel GR, Kelm M, Hendgen-Cotta U, Rassaf T. Filtration of Macrophage Migration Inhibitory Factor (MIF) in Patients with End Stage Renal Disease Undergoing Hemodialysis. PLoS One. 2015 Oct 20;10(10):e0140215. doi: 10.1371/journal.pone.0140215. eCollection 2015. PMID 26485680